CLINICAL TRIAL: NCT06821841
Title: Using Psychological Theory to Promote Physical Activity Among Peri- and Post-menopausal Working Women: A Pilot Randomised-Controlled Trial (RCT).
Brief Title: Pilot Trial of an Online Physical Activity Intervention for Peri- and Post-menopausal Working Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETH2425-0016
Record Dates: First submitted 2025-02-11; First posted 2025-02-12 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Perimenopausal Women; Postmenopausal
Keywords: online physical activity group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Physical Activity Group (Experimental)
  Interventions: Behavioral: Online Physical Activity Group; Behavioral: Information Leaflet
- Control - Information Leaflet Only (Other)
  Interventions: Behavioral: Information Leaflet

INTERVENTIONS:
Behavioral: Online Physical Activity Group — The online physical activity group will consist of four 45-60-minute sessions, which participants allocated to this group will be asked to commit to. These sessions will be delivered online and occur for 4 weeks. Discussions within the sessions will incorporate motivational interviewing, focussing on the benefits of physical activity, current physical activity levels, barriers to physical activity and overcoming these, motivation to complete physical activity, and goal setting. Participants allocated to this group will receive weekly reminders to promote attendance. Participants will also be asked to complete a weekly physical activity log that includes detail about the type of physical activity they completed, the duration, intensity, context and comments.
  Arms: Online Physical Activity Group
Behavioral: Information Leaflet — Participants will receive an information leaflet that includes information about menopause (e.g. definition, symptoms), the benefits of physical activity for menopause, recommended weekly physical activity levels (based on CMO guidelines), examples of physical activity, and signposting to online resources. Participants will be able to use the information leaflet as they wish, and complete a weekly physical activity log that includes detail about the type of physical activity completed, the duration, intensity, context and comments.

SUMMARY:
It is the purpose of this clinical trial to examine the feasibility and acceptability of a brief online physical activity group (incorporating motivational interviewing) for UK women who are currently experiencing peri- or post-menopausal symptoms and working full-time. To measure feasibility and acceptability, the following will be examined: 1. The ease that participants were recruited; 2. The proportion of participants that remained in the online physical activity group (attending at least half of the sessions); 3. The proportion of participants that remained in the study; 4. How acceptable the participants find the online physical activity group; 5. Whether there is a preliminary indications that the online physical activity group may increase participant activity levels. Once provided informed consent, all participants will be randomly allocated into either the online physical activity group (intervention arm) or the control group. Participants will be asked to complete outcome measures at the same four timepoints, as well as completing a weekly physical activity log.

DETAILED DESCRIPTION:
This pilot RCT seeks to examine the feasibility and acceptability of an online physical activity group (incorporating motivational interviewing) for UK women experiencing peri- or post-menopausal symptoms and currently working full-time. Having provided informed consent, all participants will be randomly allocated to either the online physical activity group (intervention arm) or control group. Those in the online physical activity group will be invited to attend 4-weekly sessions that last 45-60 minutes, as well as receiving and information leaflet based on Chief Medical Officer (CMO) guidelines. The control group will receive the same information leaflet based on CMO guidelines only and will be able to use this as they wish. Self-report questionnaires will be administered online at the same four timepoints; 1. Baseline (week 0-1) - all participants will complete demographic information, IPAQ, MRS and WPAI; 2. 1-week (week 1) - all participants will complete the IPAQ only; 3. Post-intervention (week 8-9) - all participants will complete the IPAQ, MRS and WPAI. Participants in the intervention arm will complete an additional feedback questionnaire; 4. 1-month follow-up (week 12-13) - all participants will complete the IPAQ, MRS and WPAI. Feasibility and acceptability will be examined by: 1. The ease that participants were recruited; 2. The proportion of participants that remained in the online physical activity group (attending at least half of the sessions); 3. The proportion of participants that remained in the study; 4. How acceptable the participants find the online physical activity group; 5. Whether there is a preliminary indications that the online physical activity group may increase participant activity levels. These outcomes will be examined against pre-defined progression criteria (based on previous literature and outlined in the outcome measures section), to determine whether the intervention is feasible and acceptable to progress to a full-scale RCT at a later date.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 30-60 years
* Currently working full-time (approximately 35+ hours per week)
* Currently experiencing perimenopausal (women with newly inconsistent menstrual cycles, >1 year since last cycle) or post-menopausal (cessation of menstrual cycle for >12 months) symptoms, which are impacting functioning
* Currently physically inactive or not meeting recommended government guidelines (150-minutes of moderate-vigorous physical activity per week)
* No comorbid health conditions that impact ability to participate in physical activity

Exclusion Criteria:

- Those who do not meet the inclusion criteria.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited to the study | 9 months from the start of recruitment
  The number of participants recruited will be compared to pre-defined progression criteria, based on existing literature, to examine the feasibility of recruitment. This progression criteria will follow a traffic light system; Green = 40-50 participants, Amber = >24 participants, Red = <24 participants.
Retention rate of participants attending the online intervention | Week 0 to 8-9
  The proportion of participants who attend at least half of the online physical activity group sessions, which will be compared to progression criteria; Green = >50%, Amber = 25-49%, Red = <25%.
The retention rate of participants who remain in the study as a whole | Week 0 to 12-13
  The proportion of participants who remain in the study, compared to progression criteria: Green = >50%, Amber = 25-49%, Red = <25%
Acceptability of the online physical activity group intervention | Week 8-9
  Participant responses to the feedback questionnaire, including Likert-scale questions and content analysis of qualitative questions. This will be compared to progression criteria; Green = High satisfaction/acceptability from the majority of participants, with a mean of 7/10 on the Likert-scale questions, Amber = Moderate/Inconsistent satisfaction and acceptability indicated, Red = Low satisfaction/acceptability from the majority of participants
Preliminary indicator of effectiveness for the primary outcome (physical activity) | Week 8-9 and 12-13
  Estimate of the between group effect size for the online physical activity group compared to control group on the International Physical Activity Questionnaire-Short Form (IPAQ-SF), from baseline [Week 0 - 1] to post-intervention and follow-up [Week 8-9 and Week 12-13, respectively]. This will be compared to progression criteria; Green = the between-group effect size is in favour of the intervention, with a substantial number of participants (>50%) showing reliable change (according to the calculated Reliable Change index; Jacobson & Truax, 1991), Amber = between-group effect size is in favour of the intervention arm, with a small number of participants showing reliable change (25-49%), Red = between-group effect size is in favour of the control group, with a minimal number of participants in the intervention group showing reliable change (<25%).

SECONDARY OUTCOMES:
Estimate of between group effect size for change on the International Physical Activity Questionnaire-Short Form (IPAQ-SF) from baseline to post-intervention and 1-month follow-up | Week 8-9 and 12-13
  Estimate of the between group effect size of the online physical activity group compared to control group on change on the International Physical Activity Questionnaire - Short Form (IPAQ-SF) from baseline (week 0-1) to post intervention (week 8-9) and follow-up (week 12-13). The IPAQ-SF is a 7-item questionnaire that assesses an individual's physical activity levels (e.g. walking, moderate-intensity, vigorous-intensity) and sedentary behaviour (e.g. sitting). Higher scores on the IPAQ-SF indicates more physical activity.
Estimate of between group effect size for the Menopause Rating Scale (MRS) from baseline to post-intervention and 1-month follow-up | Week 8-9 and 12-13
  Estimate of the between group effect size of the online physical activity group compared to control group on change on the Menopause Rating Scale (MRS) from baseline (week 0-1) to post-intervention (week 8-9) and follow-up (week 12-13). The MRS is an 11-item questionnaire that assesses the severity of various menopausal symptoms (somatic, psychological and urogenital) using a 5-point Likert-scale. Higher scores on the MRS indicate greater symptoms severity.
Estimate of between group effect size for the Work Productivity and Activity Impairment Questionnaire (WPAI) from baseline to post-intervention and 1-month follow-up | Week 8-9 and 12-13
  Estimate of the between group effect size of the online physical activity group compared to control group on the change on the Work Productivity and Activity Impairment Questionnaire (WPAI) from baseline (week 0-1) to post-intervention (week 8-9) and follow-up (week 12-13). The WPAI is a self-report questionnaire that measures the impact of a specific health difficulty on work (e.g. absenteeism, work productivity) and daily activities (e.g. household chores, hobbies). Higher scores on the WPAI indicate greater impact on work.

OTHER OUTCOMES:
Test-Retest Reliability of the International Physical Activity Questionnaire-Short Form (IPAQ-SF) | Week 0-1 (baseline) to week 1-2
  Before the intervention begins, the IPAQ-SF will be completed at baseline (week 0-1) and 1-week later. This will enable a reliability coefficient for the IPAQ-SF to be calculated for this population, which will later be used to calculate the Reliable Change Index (RCI) for participants.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Fergal Jones, Study Chair — Canterbury Christ Church University
Locations (1):
- Salomons Institute for Applied Psychology, Canterbury Christ Church University, Royal Tunbridge Wells, Kent, United Kingdom